CLINICAL TRIAL: NCT05079269
Title: Effect of Pre-operative Intravenous Crystalloids on Post-Induction Blood Pressure
Brief Title: Pre-op Fluid Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21
Record Dates: First submitted 2021-10-01; First posted 2021-10-15 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-04

CONDITIONS: Hypotension Drug-Induced; Anesthesia
Keywords: Postinduction hypotension; Perioperative fluid management
MeSH Terms: conditions — Hypotension | interventions — Crystalloid Solutions

STUDY DESIGN:
Intervention Model Description: A randomized intervention cohort study of two preoperative fluid management strategies
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The investigators will start a balanced crystalloid solution (in detail we will administer 500ml if the actual body weight is ≤90 kg: the investigators will administer 1000 ml if the actual body weight is >90 kg:) within 60 +/- 15 minutes before induction of anesthesia in the pre-operative area or at the ward, as appropriate.
  Interventions: Other: Crystalloid Solutions
- Control (No Intervention): Patients will receive the balanced crystalloid solution according to the current clinical standard of care.

INTERVENTIONS:
Other: Crystalloid Solutions — As above
  Arms: Intervention

SUMMARY:
Theoretical framework:

Hypotension during surgery directly impacts patients' postoperative outcomes and complications. Decrease in blood pressure measurements secondary to anesthetic drugs is an expected scenario in most surgical cases. Moreover, hypovolemia secondary to fast pre-operative period may facilitate post-induction hypotension which can be compensated by fluid bolus pre-operatively.

DETAILED DESCRIPTION:
Objectives:

The purpose of the study is to conduct a randomized intervention cohort study using pre-operative fluid therapy to assess its effect on blood pressure during the post-induction period. The investigators are testing the hypothesis that preoperative Crystalloid bolus decreases the risk of post-induction hypotension, specifically the time-weighted average (TWA) mean arterial pressure (MAP) under 65 mmHg during the first 20 minutes after anaesthetic induction or until surgical incision, whichever is first, compared to standard of care, which is minimal fluid administration in the pre-operative period.

Methods:

The investigators will conduct a randomized intervention cohort study using pre-operative fluid therapy to assess its effect on blood pressure during the post-induction period. The intervention group will receive a bolus of a balanced crystalloid solution within 60 ± 15 minutes before induction of anaesthesia. The control group will be treated according to the current clinical standard of care. The investigators will compare the time-weighted average (TWA) mean arterial pressure (MAP) under 65 mmHg during the first 20 minutes after anaesthetic induction or until surgical incision (whichever comes first).

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for major non-cardiac surgery
2. Having general anaesthesia
3. Are designated ASA physical status ≥2 (ranging from mild systemic disease through severe systemic disease that is a constant threat to life)
4. Subject to at least one of the following risk factors:

   1. Age ≥ 65 years
   2. History of peripheral arterial surgery
   3. History of coronary artery disease
   4. History of stroke or transient ischemic attack
   5. Serum creatinine >175 µmol/L (>2.0 mg/dl)
   6. Diabetes requiring medication
   7. Current smoking or 15 pack-year history of smoking tobacco
   8. Preoperative high-sensitivity troponin T >14 ng/L or troponin I equivalent, defined as ≥15 ng/L (Abbott assay),75 19 ng/L (Siemens assay, [Borges, unpublished]), or 25% of the 99% percentile for other assays;
   9. B-type natriuretic protein (BNP) ≥ 80 ng/L or N-terminal B-type natriuretic protein (NT-ProBNP) ≥ 200 ng/L.76,77
   10. History of atrial fibrillation
   11. Chronically taking at least one anti-hypertensive medication

Exclusion Criteria:

1. Are scheduled for carotid artery surgery
2. Are scheduled for intracranial surgery
3. Are scheduled for pheochromocytoma surgery
4. Require preoperative intravenous vasoactive medications
5. Active decompensated congestive heart failure (documented EF < 30%)
6. Chronic Kidney Disease (eGFR< 30 mL/min)
7. History of organ transplantation
8. Rectal surgical procedures
9. Patients receiving preoperative bowel preparation
10. Severe pulmonary edema

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Post-induction MAP | 60 +/- 15 minutes before induction of anesthesia until the first 20 minutes after anesthetic induction or until surgical incision (whichever comes first)
  Post-induction hypotension is defined as TWA MAP under 65 mmHg during post-induction period. We will use non-invasive continuous arterial blood pressure monitoring as feasible.
  Anesthesia staff and nurses will be blinded, and standard of care will be provided. Data from the monitor will be recorded in the anesthesia record. We will be using standard intraoperative patient monitoring system. This system will measure 3 lead ECG (electrocardiogram), SpO2 (Arterial oxygen saturation), and number of respirations continuously. The primary outcome will be the TWA MAP under 65 mmHg during the post-induction period.

SECONDARY OUTCOMES:
Vasopressors | 60 +/- 15 minutes before induction of anesthesia until the first 20 minutes after anesthetic induction or until surgical incision (whichever comes first)
  The major outcome for the vasopressor requirement will be a binary variable representing the use of vasopressors during the post-induction period. Additionally, we will compare the amount of vasopressors between the groups.
Cardiac Output (CO) | 60 +/- 15 minutes before induction of anesthesia until the first 20 minutes after anesthetic induction or until surgical incision (whichever comes first)
  The major outcome for the non-invasively measured CO will be a continuous measurement throughout pre-induction, induction of anesthesia and post-induction as feasible.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kurz, Prof, Principal Investigator — Medical University of Graz, Austria
Locations (2):
- Austria (2):
  - Medical University Graz, Graz, Styria
  - Medical University Vienna, Vienna, Vienna

IPD SHARING:
Plan to Share IPD: Yes
For electronic data management we will use the CLINCASE software (Quadratek, Berlin, Germany). Data storage and back up will be provided by IT Systems & Communications (ITSC) - IT4Science (Medical University of Vienna). Access to data is strictly controlled and will only be provided to the Sponsor (Medical University of Graz and the Medical University of Vienna), the study investigators and the ethic commission (Ethic commission of the Medical University of Vienna).
  All entries and changes in the CLINCASE software will be tracked.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be transferred immediately after patient's enrolment and will be available until the end of the study for both sponsors (Medical University of Graz, Medical University of Vienna)
Access Criteria: Access will only be provided to the Sponsor (Medical University of Graz and the Medical University of Vienna), the study investigators and the ethic commission (Ethic commission of the Medical University of Vienna).